CLINICAL TRIAL: NCT01387152
Title: Prognosis of Very Low Dose Stress First Myocardial Perfusion SPECT in Patients With Chest Pain Using an Alcyone Camera
Brief Title: Prognosis of Very Low Dose SPECT
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Andrew J. Einstein, MD, PhD, Associate Professor of Medicine, Radiology, Columbia University
Other Study IDs: AAAI0383; 10-MYO-003 (Other Grant/Funding Number: GE Healthcare)
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Chest Pain
Keywords: chest pain; myocardial perfusion scintigraphy; nuclear stress testing; low radiation dose
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Very low dose stress test protocol: Patients admitted to New York Presbyterian Hospital (NYPH)-Columbia University Medical Center with chest pain but normal or nondiagnostic electrocardiograms and at least 3 negative troponins taken 4 or more hours apart, and undergo exercise or pharmacologic stress testing using a very low dose (<6 mCi) of Tc99m tetrofosmin or sestamibi with imaging performed using acquisitions with an Alcyone camera.

SUMMARY:
Nuclear stress testing evaluates whether the heart receives enough blood, by injection of a nuclear isotope during a stress on the heart that permits taking pictures of the heart muscle. A low-radiation-dose protocol for nuclear stress testing involves injecting less of the nuclear isotope than standard protocols, by utilizing a new, more efficient camera (called an Alcyone camera) which could decrease radiation dose to patients while still providing excellent clinical information. Subjects will undergo imaging under the Alcyone camera after undergoing stress testing with exercise or a standard medication simulating exercise, and then at rest if needed. Subjects will have follow-up to measure events occurring after the test, such as death, heart attack, unstable angina, repeat emergency department visit for chest pain evaluation, or repeat imaging needed to evaluation for coronary artery disease. Radiation doses and quality of the images from the imaging with the new protocol will be recorded to compare to those used in standard nuclear imaging protocols. The primary study hypothesis is that greater than 90% of patients who have a normal very low dose stress first myocardial perfusion scintigraphy (MPS) will be free at 3 months after study of death, nonfatal myocardial infarction, unstable angina, and repeat emergency department visit for chest pain evaluation or repeat anatomical or functional cardiac imaging.

DETAILED DESCRIPTION:
See brief summary above.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with chest pain but normal or nondiagnostic electrocardiograms and at least 3 negative troponin levels taken 4 or more hours apart.
* Age greater than 18 years.
* Written informed consent is obtained by a study investigator.

Exclusion Criteria:

* Previous Myocardial perfusion scintigraphy (MPS) with evidence of scar
* Previous MPS with evidence of ischemia and no subsequent revascularization
* Known dilated left ventricle
* Known cardiomyopathy
* High pre-test probability of a perfusion defect on MPS
* Body mass index greater than 35
* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be patients who have presented to NYPH- Columbia University Medical Center with chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients free of composite endpoint | 3 months after MPS and hospital discharge (an expected average of 12 hours after MPS)
  Composite endpoint consists of:
  * death
  * non-fatal myocardial infarction
  * unstable angina
  * repeat emergency department visit for chest pain evaluation,or repeat anatomical or functional cardiac imaging

SECONDARY OUTCOMES:
Percentage of patients for whom rest imaging is needed. | 12 months after MPS and hospital discharge (an expected average of 12 hours after MPS)
Image quality on a 5 point scale | Up to 12 months after MPS and hospital discharge (an expected average of 12 hours after MPS)
  Imagine quality is assessed by 2 readers and is scored on a 5-point scale: excellent, very good, good, fair, poor.
Average effective dose of radiation received by all patients. | Up to 12 months after MPS and hospital discharge (an expected average of 12 hours after MPS)
Average effective dose received by patients for whom stress-only MPS is performed. | Up to 12 months after MPS and hospital discharge (an expected average of 12 hours after MPS)
Duration of stress test | Up to 12 months after MPS and hospital discharge (an expected average of 12 hours after MPS)
Duration of hospitalization | Up to 12 months after MPS and hospital discharge (an expected average of 12 hours after MPS)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Einstein, MD, PhD, Principal Investigator — NYPH- Columbia University Medical Center
Locations (1):
- New York Presbyterian Hospital- Columbia University Medical Center, New York, New York, United States